CLINICAL TRIAL: NCT06944756
Title: Effects of Global Postural Reeducation Compared to Scapular Stabilization Exercises on Pain, Flexibility, and Function of Patients With Shoulder Pain Associated With Scapular Dyskinesia
Brief Title: Effects of Global Postural Reeducation Versus Scapular Stabilization Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCR&AHS/REC/MS-OMPT/S19/013
Record Dates: First submitted 2025-04-07; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Scapular Dyskinesis
Keywords: Scapular Dyskinesia; Shoulder Pain; Global Posture Reeducation
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and assessor blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A: GPR (Experimental): Two stretching postures were maintained for 10 minutes each.
  Interventions: Other: Global Postural Reeducation
- GROUP B: SSE (Experimental): 1) Push up plus and 2) press up, were selected in reference to a study for scapular stabilization.
  Interventions: Other: Scapular Stabilization Exercises

INTERVENTIONS:
Other: Global Postural Reeducation — Two stretching postures were maintained for 10 minutes each.
  * In order to stretch the posterior muscle chain(the supine posture with hip ﬂexion, which stretches the posterior muscle chain) the patient lay in the supine position with the occipital, lumbar, and sacral spine stabilized, with the lower limbs at 90° hip flexion, and performed gradual knee extensions, and dorsiﬂexion of the ankle.
  * In order to stretch the anterior muscle chain (the supine posture with leg extension, which progressively stretches the anterior muscle chain) the patient lay in the supine position with the upper limbs abducted at 30° and the forearms supine.. Hips were flexed, abducted, and laterally rotated, with the soles of the feet touching each other. Gradually, respecting the patient's limits, the lower limbs were extended as much as possible and adduction of the upper limbs.
  Arms: GROUP A: GPR
Other: Scapular Stabilization Exercises — 1) Push up plus and 2) press up, were selected in reference to a study for scapular stabilization.
  During the 5-week intervention training, sets of repetitions were increased progressively. In the ﬁrst week participants performed 3 sets of each exercise (10 repetitions × 10-second duration each) and worked up to a maximum of 5 sets of 10 repetitions in the last weeks of the intervention.
  Arms: GROUP B: SSE

SUMMARY:
Shoulder pain is an experience that most of the people can expect to deal in their lives due to over-exertion or postural asymmetries, which may or may not have it interfering with the normal activities of their daily living. Shoulder pain associated with scapular dyskinesia can be associated with restricted joint range of motion and loss of muscle strength, and is among the most common conditions treated by physical therapists. The patho-mechanisms of shoulder pain are only scarcely known but it is associated with both psychosocial and physical factors. Although there is some evidence of pain reduction, improving range of motion and function occurring following global posture reeducation, scapular stabilizing exercise, it is not known how the training influences the muscle activities of persons shoulder pain associated scapular dyskinesia.

DETAILED DESCRIPTION:
The objective of this study will be to compare the effects of Global Postural Reeducation and Scapular Stabilization Exercises on pain, range of motion, and activity restriction in patient with shoulder Pain. Data will be collected from Hajra complex and Riphah Rehabilitation center Lahore. A sample of 30 patients will be included and divided into two group. One group will receive Global Postural Reeducation and other group will receive Scapular Stabilization Exercises. All subjects will receive a total of ten treatment sessions twice a week over the period of 5 weeks lasting for 40 minutes. Outcome will be measured with Goniometer, NPRS, DASH/PSS. The data will be analyse using SPSS v 25. The normality of the data will be assessed by Shapiro-Wilks test of normality and uniformity, based on which parametric or non-parametric test will be applied to determine within the group and across the group difference in two groups. Independent sample T test / Mann Whitney U test will be applied to determine any significant difference across the two groups. Repeated Measure ANOVA / Friedman ANOVA will be used to determine any significant difference with in each treatment group. A difference with p value less than 0.05 will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders.
* SD of type I with scapular malposition, inferior medial border prominence, coracoid pain and malposition, and dyskinesia of scapular movement (SICK) Scapula Rating Scale, in association to shoulder pain (pain for at least 3 months).
* Pain intensity ranges from 2-9 on scale of shoulder in last month.

Exclusion Criteria:

* Additional cervical or shoulder pathology (cervical stenosis, myelopathy, prolapsed intervertebral disk )
* Pre-diagnosed winged scapula due to lesions of the long thoracic nerve or spinal accessory nerve.
* Patients with shoulder instability
* Medical red flag history (tumor, metabolic diseases, rheumatoid arthritis, osteoporosis or Infection)
* Any Neurological disorder that affects shoulder
* History of Severe trauma or any fracture of shoulder girdle
* Hypertension (Systolic BP[160, diastolic BP[100])
* Cardiovascular diseases (e.g., chest pain during physical exercise, heart failure, myocardial infarction)
* Postoperative conditions in the neck and affected shoulder region Pregnancy

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-06 (Actual); Primary Completion 2019-07-06 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Shoulder Flexion Range of Motion | Pre, 3rd week, 5th week
  Goniometer
Shoulder Abduction ROM | Pre, 3rd week, 5th week measured using degree of movement (160 to 180)
  Goniometer
Shoulder Pain | Pre, 3rd week, 5th week (Score measuring on on a scale of 0 to 10, 0 being no Pain and 10 being worst)
  Numeric Pain Rating Scale
Shoulder Disability | Pre, 3rd week, 5th week (scoring 0-100, 0 being no disability and 100 being most sever disability)
  Disability of arm shoulder and hand
Shoulder Function | Pre, 3rd week, 5th week (scoring 0-100, 0 being poor shoulder function and 100 being most best shoulder fucntions)
  Pennsylvania Shoulder scale

CONTACTS AND LOCATIONS:
Overall Officials: Aiza Yousaf, DPT, Principal Investigator — Riphah International University
Locations (1):
- Ali Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No